CLINICAL TRIAL: NCT06669052
Title: Liposomal Iron 30 mg Supplement in Non-anemic Pregnant Females an Observational Study
Brief Title: Liposomal Iron 30 mg Supplement in Non-anemic Pregnant Females
Acronym: LITSNPF
Status: Not yet recruiting | Type: Observational
Sponsor: Orchidia pharmaceutical Industries (Industry)
Collaborators: MARS-Global (Other)
Responsible Party: Sponsor
Other Study IDs: 00012098
Record Dates: First submitted 2024-10-28; First posted 2024-11-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Anemia of Pregnancy; Iron Deficiency Anemia
Keywords: 30 mg liposomal irom; non-anemic pregnant females; observational study; hemoglobin level; Second trimester
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — Capsules

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1 arm group, pregnant non-anemic females, second trimester.: Liposomal iron, capsules, 1 Capsule with food or few hours before or after taking other medication once daily. 1 arm group, Participants in this study will receive a daily oral dose of 30 mg Iron for a duration of 90 days. The liposomal formulation is designed to enhance the bioavailability of iron, potentially reducing gastrointestinal side effects.
  Interventions: Dietary Supplement: 30 mg liposomal iron, capsules

INTERVENTIONS:
Dietary Supplement: 30 mg liposomal iron, capsules — a dietary supplement capsule, of mainly 30 mg liposomal iron, and Vitamin C 70mg, vitamin D3 400IU, vitamin B6 1.75 mcg, Folate 1000 mcg, b=vitamin B12 10 mcg. all in capsulated in 1 Hard gelatin capsule

SUMMARY:
Protocol Summary: Liposomal Iron Supplementation in Non-anemic Pregnant Females This observational study aims to evaluate the efficacy and safety of daily liposomal iron supplementation (30 mg) in non-anemic pregnant women during their second trimester of pregnancy. The study will focus on pregnant females aged 18-45 years with low-risk, singleton pregnancies who are non-anemic (hemoglobin ≥10.5) at 14-16 weeks gestation.

Primary Research Question:

Does daily supplementation with 30 mg liposomal iron effectively maintain maternal hemoglobin levels over 90 days? Measured by: The difference in maternal hemoglobin levels between baseline and after 90 days of treatment in women recruited at 14-16 weeks gestation.

Secondary Research Questions:

What are the effects of liposomal iron supplementation on serum ferritin levels? Measured by: Changes in serum ferritin levels between baseline and after 90 days of treatment.

What is the safety profile of liposomal iron supplementation during pregnancy? Measured by: Maternal gastrointestinal side effects monitored at each prenatal visit (day 30, 60, and 90).

What is the compliance rate with liposomal iron supplementation? Measured by: Participant-reported compliance assessed at each prenatal visit (day 30, 60, and 90).

Participants will:

Receive daily liposomal iron supplementation (30 mg) for 90 days. Attend regular prenatal visits for monitoring at days 30, 60, and 90. Complete questionnaires about compliance and any adverse effects at each visit. Undergo blood tests to measure hemoglobin and serum ferritin levels at baseline and day 90.

This multi-center study will involve 714 participants across 100 sites, with recruitment beginning in November 2024 and study completion expected by July 2025. The study's findings will contribute to understanding the role of liposomal iron supplementation in preventing iron deficiency during pregnancy and its potential advantages over traditional iron supplements in terms of tolerability and compliance.

DETAILED DESCRIPTION:
This observational, prospective study aims to evaluate the safety and efficacy of Liposomal Iron 30 mg supplement in non-anemic pregnant women during the second trimester (gestational weeks 14 to 16). Conducted at approximately 100investigative sites across Egypt, the study targets the enrollment of 714 participants.

The primary objective is to assess the impact of daily supplementation with liposomal iron over a 90-day period on maternal health. The study will monitor participants through routine prenatal visits, where data on adverse effects will be collected alongside routine hemoglobin and serum ferritin measurements.

The study will utilize a Data and Safety Monitoring Board (DSMB) to ensure oversight of participant safety and the integrity of study data. The DSMB will regularly review safety information and study progress, providing recommendations to the sponsor regarding the continuation or termination of the trial if necessary.

Statistical analyses will be performed using methods appropriate for the data collected, ensuring that the results will robustly assess the safety and efficacy of the liposomal iron supplement.

This study is designed to provide critical insights into iron supplementation for pregnant women, addressing a significant public health issue by exploring a formulation that may enhance compliance and reduce gastrointestinal side effects associated with traditional iron supplements.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant females; gestational age from 14 to 16 weeks Age 18-45 years
* Low-risk pregnancy is defined as a pregnancy in which there is no high risk of problems or unfavorable outcomes, and the expectant mother and fetus are typically healthy
* Non-anemic women at the time of recruitment (hemoglobin level not less than 10.5. Hemoglobin measured within 2 or 3 weeks of recruitment
* Singleton pregnancy
* Agree to participate in the study including data collection from medical records and participation in related questionnaires.

Exclusion Criteria:

* Inadequate medical records
* Pregnant women living in areas away from the recruitment center
* Had any chronic health problem.
* Women with any form of hereditary anemia including sickle cell anemia, thalassemia, and Glucose-6-phosphate dehydrogenase (G6PD) deficiency.
* History of antepartum bleeding
* Refuse to sign the informed consent.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant non-anemic females
Study Population: This study will include non-anemic pregnant females > 18 years old taking liposomal iron in non-anemic pregnant females as an iron supplement during 14-16 weeks of pregnancy. The study will be conducted at approximately 100 investigative sites in Egypt. Recruitment will stop when approximately 714 subjects are enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 714 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Measure the change in Maternal Hemoglobin Level | Baseline and after 90 days of treatment
  Measurement: To assess the efficacy of liposomal iron 30 mg once daily on hemoglobin levels in non-anemic pregnant females, measurement: Hemoglobin (g/dL)

SECONDARY OUTCOMES:
Measures change in Serum Ferritin Levels to evaluate changes in serum ferritin levels following liposomal iron supplementation. | Baseline and after 90 days of treatment
  Measurement: Ferritin (µg/L)
Assessment of Maternal Gastrointestinal Side Effects, to monitor gastrointestinal side effects associated with liposomal iron supplementation during pregnancy. | Days 30, 60, and 90 of treatment
  Measurement: Incidence of side effects (Count of reported instances)
Compliance Rate with Supplementation, to assess patient compliance with liposomal iron supplementation. | At each prenatal visit (Days 30, 60, and 90)
  Measurement: Compliance rate (Percentage)

CONTACTS AND LOCATIONS:
Overall Officials: Yasser S El Kassar, Prof. Dr., Principal Investigator — Faculty of medicine Alexandria university, obstetrics and gynecology department

IPD SHARING:
Plan to Share IPD: Undecided
Currently, it is undecided whether individual participant data (IPD) collected in this study will be shared with other researchers. This decision will be evaluated upon the study's completion